CLINICAL TRIAL: NCT07057375
Title: A Prospective Randomized Study to Investigate the Effect of Pulsed Electromagnetic Field Therapy on Muscle Mass and Muscle Strength in Prostate Cancer Patients Treated With Androgen Deprivation Therapy
Brief Title: The Effect of Pulsed Electromagnetic Field Therapy on Muscle Mass and Muscle Strength in Prostate Cancer Patients Treated With Androgen Deprivation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Chi Fai, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CRE-2024.600-T
Record Dates: First submitted 2025-05-04; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: ADT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Therapy (Active Comparator): Pulsed electromagnetic fields therapy will be delivered using the BIXEPS system (QuantumTX, Singapore).
  Interventions: Device: Pulsed electromagnetic fields Thearpy
- Sham Therapy (Sham Comparator): Sham thearpy will be delivered using the BIXEPS system (QuantumTX, Singapore).
  Interventions: Device: Sham Therapy

INTERVENTIONS:
Device: Pulsed electromagnetic fields Thearpy — Pulsed electromagnetic fields (PEMF) is a non-invasive and non-thermal treatment used to stimulate muscle regeneration, resulting in increased muscle mass and strength.
  Arms: Active Therapy
Device: Sham Therapy — Sham Therapy
  Arms: Sham Therapy

SUMMARY:
This study is to assess the effect of Pulsed electromagnetic fields (PEMF) on improving muscle mass and strength in prostate cancer patients with ADT.

DETAILED DESCRIPTION:
This randomised parallel-group study assesses the efficacy, safety and tolerability of Pulsed electromagnetic fields (PEMF) on the muscle mass and strength in PCa patients treated with ADT.Treatment will be delivered using the BIXEPS system (QuantumTX, Singapore). During each treatment, the subject's quadriceps (thigh) region will be put into the machine and treated for 10 minutes for each lower limbs. The whole treatment consists of 1 therapy session per week for 12 weeks. The two lower limbs will be treated alternatively during the treatment. A set of assessments, including body composition assessment, muscle function assessment, questionnaire assessment, and blood and urine for inflammation and cytokines measurement, will be performed at baseline before the start of the first treatment, week 5 and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with age greater than or equal to 18 years old.
* Histologically documented PCa
* No evidence of distant metastasis (M1 disease)
* With ADT exposure from six months to three years
* Expected to continue for at least six months
* At least four weeks after radical prostatectomy or completed radiotherapy

Exclusion Criteria:

* Patients are still under active treatment, such as radiotherapy
* Patients who are unable to walk for 400 m or undertake exercise that will affect the clinical assessment of muscle strength
* Patients with amputated lower limbs or other body deformities that will affect the treatment protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Time Up and Go tests (TUG test) | Baseline, Week 5, Week 12
  Changes in time for Time Up and Go tests (TUG test) at the end of the 12-week treatment

SECONDARY OUTCOMES:
Appendicular skeletal muscle mass | Baseline, Week 5, Week 12
  Changes in appendicular skeletal muscle mass at the end of the 12-week treatment
Body Mass Index (BMI) | Baseline, Week 5, Week 12
  Changes in BMI at the end of the 12-week treatment
Calf circumference | Baseline, Week 5, Week 12
  Changes in calf circumference at the end of the 12-week treatment
Hand grip Strength | Baseline, Week 5, Week 12
  Changes in hand grip strength at the end of the 12-week treatment
Five times sit-to-stand tests | Baseline, Week 5, Week 12
  Changes in time for Five times sit-to-stand tests at the end of the 12-week treatment
Quality of life measured by 5-level EQ-5D version (ED-5Q-5L)questionnaire | Baseline, Week 5, Week 12
  Quality of life measured by ED-5Q-5L questionnaire, which include the the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS range from 0 to 100).the higher the score the better in quality of life
Sarcopenia measured by SARC-F(strength, walking, rising from a chair, climbing stairs, and experiencing falls) score | Baseline, Week 5, Week 12
  Changes in SARC-F scores at the end of the 12-week treatment. The score equal to or greater than 4 is predictive of sarcopenia
Concentration of Cytokines and inflammatory markers | Baseline, Week 5, Week 12
  Changes in a panel of cytokines and inflammatory markers at the end of 12 week treatment
Quality of life measured by FACT-P Questionnaire | Baseline, Week 5, Week 12
  The higher the score, the better of Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith MR, Saad F, Egerdie B, Sieber PR, Tammela TL, Ke C, Leder BZ, Goessl C. Sarcopenia during androgen-deprivation therapy for prostate cancer. J Clin Oncol. 2012 Sep 10;30(26):3271-6. doi: 10.1200/JCO.2011.38.8850. Epub 2012 May 29. PMID 22649143
- [Background] Basaria S, Lieb J 2nd, Tang AM, DeWeese T, Carducci M, Eisenberger M, Dobs AS. Long-term effects of androgen deprivation therapy in prostate cancer patients. Clin Endocrinol (Oxf). 2002 Jun;56(6):779-86. doi: 10.1046/j.1365-2265.2002.01551.x. PMID 12072048
- [Background] Beaudart C, McCloskey E, Bruyere O, Cesari M, Rolland Y, Rizzoli R, Araujo de Carvalho I, Amuthavalli Thiyagarajan J, Bautmans I, Bertiere MC, Brandi ML, Al-Daghri NM, Burlet N, Cavalier E, Cerreta F, Cherubini A, Fielding R, Gielen E, Landi F, Petermans J, Reginster JY, Visser M, Kanis J, Cooper C. Sarcopenia in daily practice: assessment and management. BMC Geriatr. 2016 Oct 5;16(1):170. doi: 10.1186/s12877-016-0349-4. PMID 27716195
- [Background] Saylor PJ, Smith MR. Metabolic complications of androgen deprivation therapy for prostate cancer. J Urol. 2013 Jan;189(1 Suppl):S34-42; discussion S43-4. doi: 10.1016/j.juro.2012.11.017. PMID 23234628
- [Background] Greenspan SL, Coates P, Sereika SM, Nelson JB, Trump DL, Resnick NM. Bone loss after initiation of androgen deprivation therapy in patients with prostate cancer. J Clin Endocrinol Metab. 2005 Dec;90(12):6410-7. doi: 10.1210/jc.2005-0183. Epub 2005 Sep 27. PMID 16189261
- [Background] Storer TW, Magliano L, Woodhouse L, Lee ML, Dzekov C, Dzekov J, Casaburi R, Bhasin S. Testosterone dose-dependently increases maximal voluntary strength and leg power, but does not affect fatigability or specific tension. J Clin Endocrinol Metab. 2003 Apr;88(4):1478-85. doi: 10.1210/jc.2002-021231. PMID 12679426
- [Background] Galvao DA, Nosaka K, Taaffe DR, Spry N, Kristjanson LJ, McGuigan MR, Suzuki K, Yamaya K, Newton RU. Resistance training and reduction of treatment side effects in prostate cancer patients. Med Sci Sports Exerc. 2006 Dec;38(12):2045-52. doi: 10.1249/01.mss.0000233803.48691.8b. PMID 17146309
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Hanson ED, Srivatsan SR, Agrawal S, Menon KS, Delmonico MJ, Wang MQ, Hurley BF. Effects of strength training on physical function: influence of power, strength, and body composition. J Strength Cond Res. 2009 Dec;23(9):2627-37. doi: 10.1519/JSC.0b013e3181b2297b. PMID 19910811
- [Background] Denison HJ, Cooper C, Sayer AA, Robinson SM. Prevention and optimal management of sarcopenia: a review of combined exercise and nutrition interventions to improve muscle outcomes in older people. Clin Interv Aging. 2015 May 11;10:859-69. doi: 10.2147/CIA.S55842. eCollection 2015. PMID 25999704
- [Background] Esper P, Mo F, Chodak G, Sinner M, Cella D, Pienta KJ. Measuring quality of life in men with prostate cancer using the functional assessment of cancer therapy-prostate instrument. Urology. 1997 Dec;50(6):920-8. doi: 10.1016/S0090-4295(97)00459-7. PMID 9426724
- [Background] Wong CK, Choi EP, Tsu JH, Ho BS, Ng AT, Chin WY, Yiu MK. Psychometric properties of Functional Assessment of Cancer Therapy-Prostate (FACT-P) in Chinese patients with prostate cancer. Qual Life Res. 2015 Oct;24(10):2397-402. doi: 10.1007/s11136-015-0993-8. Epub 2015 Apr 16. PMID 25877953